CLINICAL TRIAL: NCT00473421
Title: "How do Contrast Medias in Bone Cement Affect DXA Measurements After THR"
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Human sementstudie
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Primary and Secondary Osteoarthritis in Hip
MeSH Terms: interventions — Barium Sulfate; zirconium oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Barium Sulphate and Zirconium Oxide

SUMMARY:
Joint replacement is a well-documented and cost effective treatment of degenerative diseases in the hip (1,2). There are two different principles of fixation of prosthesis components; cemented and uncemented. The most common mode of fixation in Scandinavia has historically been with bone cement. In the recent years a reverse hybrid combination (uncemented stem and cemented cup) is gaining popularity, especially in Norway.

Beside luxation, infection and venous thromboembolism, the problem with aseptic loosening is a known complication. A marker for aseptic loosening is local bone loss around the components. This is measured with a densiometer and the method is Dual Energy X-ray Absorbtiometry (DXA). Periprosthetic bone loss is evaluated by series of DXA scans around the components over time. This enables us to follow changes in bone mineral density (BMD) close to the prosthesis.

We want to compare cemented and uncemented prostheses with this technique. This is a problem since we don't know how much different contrast medias in bone cement affect DXA scans. This area is poorly investigated. Attempts have been made to exclude the cement-mantle from the measurements both digitally and manually, but these have showed poor precision. A kind of consensus of assuming that contrast medias in bone cement give an increase in measured BMD of 20% (4). This is used when comparing cemented and uncemented components.

We have preformed laboratory tests of different cements. Zirconium oxide (ZrO2) and Barium sulphate (BaSO4) are used as radiopacifiers. These contrast medias have different properties. Our test showed that Zirconium give 63% higher BMD when we scanned cement alone.

This is supported by a cadaver study showing significant differences between contrast free cement and ZrO2 /BaSO4 containing cements.

It is our opinion that it is necessary to perform a prospective study to investigate this more thoroughly.

The hypothesis of this study is that it is not accurate enough to add 20% in BMD for cemented implants when comparing them with uncemented implants. It is probably necessary to take into account the amount of cement used and kind of contrast medium.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis

Exclusion Criteria:

* more than 80 yrs
* systemic disease

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, MD Ph.D, Study Director — Ullevaal University Hospital; Jon Dahl, MD, Principal Investigator — Ullevaal Univerity hospital
Locations (1):
- Ullevaal university hospital, Oslo, Norway

REFERENCES:
- [Derived] Flatoy B, Dahl J, Rohrl SM, Nordsletten L. Does radiopaque cement conceal periprosthetic bone loss around femoral stems? Hip Int. 2020 Nov;30(6):731-738. doi: 10.1177/1120700019863352. Epub 2019 Jul 30. PMID 31359800